CLINICAL TRIAL: NCT05906329
Title: A Clinical Study on Low-dose Radiotherapy Combined With Conventional Fractionated Radiotherapy in Non Small Cell Lung Cancer After Immunotherapy Resistance
Brief Title: Low-dose Radiotherapy Combined With Conventional Fractionated Radiotherapy in Lung Cancer After Immunotherapy Resistance
Acronym: FL002
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Jiandong Zhang, Chief physician, Qianfoshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-KY-2023（015）
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Cancer Patients
Keywords: lung cancer, radiotherapy, immunotherapy resistance
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-dose radiotherapy combined with conventional radiotherapy after immunotherapy resistance (Other): By using enhanced CT to locate the chest, abdomen, and pelvis, the target area was delineated. The lesion was a visible lymph node with a short diameter of ≥ 1cm, and there was metastasis confirmed by two deputy chief physicians based on enhanced MR and PET/CT examination results. Select the primary lesion, the largest metastatic lesion, or the lesion causing symptoms, and perform routine segmentation (1.8-2Gy/f, 40Gy-60Gy). For the remaining lesions, at least one easily assessable and measurable lesion should be selected as the observation lesion. Unselected lesions (≤ 10) should be given 1.6Gy/f, 1f/w, 4-6 times in total. The immunotherapy plan is carried out according to the specific dose and interval of the original immune plan. Usually, immunotherapy is combined with radiotherapy at a frequency of once every 3 weeks until progression.
  Interventions: Radiation: Low-dose radiotherapy combined with conventional fractionated radiotherapy

INTERVENTIONS:
Radiation: Low-dose radiotherapy combined with conventional fractionated radiotherapy — Select the primary lesion, the largest metastatic lesion, or the lesion causing symptoms, and perform routine segmentation (1.8-2Gy/f, 40Gy-60Gy). For the remaining lesions, at least one easily assessable and measurable lesion should be selected as the observation lesion. Unselected lesions (≤ 10) should be given 1.6Gy/f, 1f/w, 4-6 times in total.

SUMMARY:
Pre-clinical and clinical studies have shown that low-dose radiation therapy has good immune regulatory effects, activates different anti-tumor immune pathways, and regulates tumor stroma to better promote T cell infiltration. Conventional fractionated radiotherapy increases antigen release and presentation, and stimulates immune cells. In theory, the combination of the two can reverse immune resistance. Our study aims to clarify the efficacy and safety of low-dose radiotherapy combined with conventional fractionated radiotherapy in reversing immune therapy resistance for patients with non-small cell lung cancer, including objective response rate (ORR), progression free survival time (PFS), disease control rate (DCR), health-related quality of life assessment (HRQoL), and incidence of adverse events (AEs).

DETAILED DESCRIPTION:
This study is a researcher initiated, prospective, single arm, open clinical study.

Patients with non-small cell lung cancer who have undergone first-line or multi-line immunotherapy and have no standard treatment option after resistance are recruited in Department of Radiotherapy in the First Affiliated Hospital of Shandong First Medical University. Patients who meet the conditions shall be treated after signing a written informed consent form. Radiotherapy localization was performed through enhanced CT, and the target area was delineated. The lesion included the primary lesion and lymph nodes with a visible short diameter of ≥ 1cm, and there was metastasis confirmed by two deputy chief physicians based on enhanced MR and PET/CT examination results.

The primary lesion, the largest metastatic lesion, or the lesion causing symptoms are selected and performed conventional fractionated radiation of 1.8-2Gy/f, 40Gy-60Gy. For the remaining lesions, at least one easily assessable and measurable lesion should be selected as the observation lesion. Unselected lesions (≤ 10) should be given 1.6Gy/f, 1f/w, 4-6 times in total.

The immunotherapy regimen is implemented according to the specific dose and interval of the original immunotherapy regimen, such as synchronous combination chemotherapy or anti angiogenic drug therapy.

Immunotherapy is combined with radiotherapy at a frequency of once every 3 weeks until progression.

The attending physician is responsible for developing personalized follow-up plans based on the patient's personal situation, daily diagnosis and treatment routines, and standards.

Evaluate the incidence of ORR, PFS, DCR, HRQoL, AE, and sAE according to the guidelines for response criteria for use in trials testing immunotherapeutics (iRECIST) to evaluate the patient's degree of benefit in this trial.

Regarding the determination of immunotherapy resistance, if the tumor does not respond to initial immunotherapy and does not respond after more than 6 weeks of exposure to immune drugs, primary resistance may occur and imaging is needed to confirm the disease progression again. If two or more deputy chief physicians evaluate and determine the disease progression, immunotherapy resistance may occur. On the other hand, if the drug exposure time is more than 6 months, the tumor does not respond, and the acquired drug resistance may occur, including the new drug-resistant mutant derived from the tumor and the changes in the tumor microenvironment. The disease progress also needs to be re determined by imaging. If the disease progress is determined after the evaluation of more than two deputy chief physicians, the immunotherapy drug resistance occurs.

The quality control of all stages of clinical trials will be strictly implemented, including relevant evaluation indicators, participants, and a complete management system will be established.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients are able to understand the informed consent form, voluntarily participate and sign the informed consent form.

  2. Age range from 18 to 65 years old, regardless of gender.

  3. ECOG level 0-1; Expected life>6 months.

  4. At least get into a liquid diet.

  5. No history of severe allergies.

  6. Hemoglobin ≥ 100 g/L, WBC ≥ 3.5 x10~9/L, neutrophils ≥ 1.8 x10~9/L, platelets ≥ 10 x10~9/L; AST and ALT ≤ 2.5 × normal upper limit, AKP ≤ 2.5 × normal upper limit.

  7. Non small cell lung cancer (adenocarcinoma, large cell carcinoma, squamous carcinoma, adenosquamous carcinoma, sarcomatoid carcinoma) confirmed by cytology or histology.

  8. Complete clinical data.

  9. ≤ 10 primary and regional metastatic lymph nodes and distant metastatic lesions, and ≤ 5 organ metastases.

  10. Malignant tumor patients with immune therapy resistance (evaluated after 6-8 weeks of treatment and no improvement in clinical symptoms) without standard treatment options.

  11. There are measurable primary lesions, regional lymph node metastasis, and distant metastatic lesions.

Exclusion Criteria:

* 1. Missing key patient information (pathological diagnosis, radiation dose, imaging examination, previous treatment plans, etc.).

  2. Refusal or lack of cooperation in research.

  3. Patients who have participated in other clinical studies/trials within three months.

  4. Patients with brain metastases.

  5. The researcher determines that there are any patients who are not suitable to participate in the study.

  6. Accompanied by severe infections.

  7. Serious liver disease (such as cirrhosis), kidney disease, respiratory disease or chronic system diseases such as uncontrollable diabetes and hypertension; Patients who cannot tolerate radiation therapy.

  8. Previous occurrence of immune related toxic side effects (immune myocarditis, pneumonia, etc.).

  9. Previous history of radiation therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-31 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR | Eighteen months
  To evaluate the objective effective rate of low-dose radiotherapy combined with conventional fractionated radiotherapy and immunotherapy in patients with non-small cell lung cancer after immunotherapy resistance without standard regimens.

SECONDARY OUTCOMES:
PFS | Eighteen months
  To evaluate the progression-free survival (PFS) of patients with advanced malignant tumors after low-dose radiotherapy combined with conventional fractionated radiotherapy and immunotherapy without standard regimens after immunotherapy resistance.
DCR | Eighteen months
  To evaluate the proportion of patients with optimal response to low-dose radiotherapy and conventional fractionated radiotherapy combined with immunotherapy to achieve complete response, partial response, or disease control after no standard regimen was available for immunotherapy resistance.
HRQoL、AE、SAE | Eighteen months
  Evaluation of health related quality of life and safety of post- low-dose radiotherapy combined with conventional fractionated radiotherapy and immunotherapy in patients with non-small cell lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Pingping Hu, Dr., Principal Investigator — Deputy chief physician
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital)16766 Jingshi Road, Jinan City, Jinan, In Shandong Province, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yin L, Xue J, Li R, Zhou L, Deng L, Chen L, Zhang Y, Li Y, Zhang X, Xiu W, Tong R, Gong Y, Huang M, Xu Y, Zhu J, Yu M, Li M, Lan J, Wang J, Mo X, Wei Y, Niedermann G, Lu Y. Effect of Low-Dose Radiation Therapy on Abscopal Responses to Hypofractionated Radiation Therapy and Anti-PD1 in Mice and Patients With Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2020 Sep 1;108(1):212-224. doi: 10.1016/j.ijrobp.2020.05.002. Epub 2020 May 15. PMID 32417411